CLINICAL TRIAL: NCT05928078
Title: A Home-based e-Health Intervention of Demanding Cognitive Exercise for the Improvement of Cardiorespiratory Fitness and Cognitive Function in the Elderly: MOVI-ageing.
Brief Title: A Home-based e-Health Intervention in the Elderly: MOVI-ageing
Acronym: MOVI-ageing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, CELIA ÁLVAREZ BUENO, Professor, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PI22/00878 PI22/00878
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will develop their usual activity
- Intervention (Experimental): Participants will use the e-Health platform
  Interventions: Behavioral: intervention

INTERVENTIONS:
Behavioral: intervention — Participants will be required to use the MOVI-ageing platform 3 times a week for 12 weeks. The platform will include videos of cognitively demanding physical activities designed and guided by health professionals, who will also be able to check compliance with the intervention.
  Arms: Intervention

SUMMARY:
This protocol study aims to evaluate the efficacy of the MOVI-ageing intervention, a complex home-based eHealth intervention of cognitive-demanding exercise for the elderly, in improving: global cognitive function and basic cognitive functions and cardiorespiratory and muscular fitness.

In addition, this sudy aims to evaluate the efficacy of the MOVI-ageing intervention, in improving: body composition (waist circumference and fat percentage), blood pressure, and health-related quality of life.

The MOVI-ageing project has been designed in three phases comprising: i) a tool development study; ii) a 12-week randomized efficacy/feasibility trial of the intervention; and iii), a large-scale implementation phase with a 12-week randomized trial.

The investigators will use a qualitative approach to improve the plataform design with the users perspective. Participants will have access to a platform where participants will be able to view videos of cognitively demanding physical exercise programs.

The videos will be directed by an avatar and the research staff will be able to know the degree of compliance with the program and the correct execution of the program through the use of Physio Galenus technology. The platform will have information on how to be more active, and chat lines to communicate with the research group. Participants will receive feedback on their compliance with the routines and reinforcement messages.

DETAILED DESCRIPTION:
This study will be carried out in three phases. During the first phase, the research team will conduct a literature review and focus groups to implement in the development of the online platform the information available in the scientific evidence and the needs and expectations of the people who will use it.

The second phase will include the implementation of the platform and its piloting in a small sample of the population. This second phase will allow the researchers to improve the platform and its access based on the results and user experiences. During the third phase the platform will be made accessible to a larger population group to show its effect on improving cognitive function and cardiorespiratory fitness in the elderly

ELIGIBILITY:
Inclusion Criteria:

* are 60 years of age or older of both genders;
* are retired regardless of the reason for retirement;
* do not meet frailty criteria according to Fried criteria;
* without disabilities for activities of daily living;
* living independently;
* without cognitive impairment as determined by the Mini-Mental test greater than 24 (considering the degree of schooling of the participants);
* able to walk at least 20 meters with or without walking aids.

Exclusion Criteria:

* mobility problem;
* serious health problem (e.g., recent myocardial infarction, recent heart attack, etc.). recent myocardial infarction, uncontrolled diabetes or uncontrolled hypertension);
* orthopedic or neurological disease that prevents training;
* Alzheimer's disease or dementia;
* progressive or terminal terminal illness;
* acute or chronic illness;
* history of heart attack;
* history of vertigo or recent head injury;
* health problems that may affect the ability to perform the EF programs (e.g. acute and painful joint inflammation, impaired mobility after a stroke), or any unstable health condition;
* use of medications that act at the neuron level (e.g., psychotropic medications);
* signs of incipient depression;
* pathology that makes it difficult to use the computer application through which the FE program will be developed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  Using the Minimental State Examination (MMSE) for global function
Change in cardiorespiratory fitness | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  6 minutes walking test (6MWT)

SECONDARY OUTCOMES:
Change in Health-related quality of life | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  SF-12 test
Change in Depression, anxiety and stress | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  Yesavage's 15-item GDS questionnaire
Change in Psychological well-being | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  Scale proposed by Ryff and translated and validated in Spanish by Diaz et al
Change in Physical activity | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  Axivity 6axes accelerometers (Axivity LTd. ) for seven consecutive days
Change in Physical function | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  Short Portable Physical Battery scale
Change in Concern about falls | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  Falls Efficacy Scale International (FES-I)
Change in Weight | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  the mean of two measurements (using a scale (Seca® 861) with the participant barefoot and lightly clothed.
Change in Height | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  the mean of two measurements with a wall-mounted stadiometer (Seca® 222), with the participant barefoot and in an upright position while the sagittal midline of the back touches the vertical bar.
Change in Body mass index (BMI) | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  as weight (kg)/height2 (m2).
Change in Waist circumference | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  the mean of three measurements using a flexible tape measure at the midpoint between the last rib and the iliac crest at the end of a normal exhalation.
Change in Body fat percentage | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  the mean of two measurements using an eight-electrode Tanita® Segmental-418 bioimpedance system (Tanita Corp.
  Tokyo, Japan).
Change in Body composition by densitometry | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  With the DXA
Change in HbA1c | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  using the ADAMS A1c HA-8180V analyzer (Menarini Diagnostics®), a method certified by the NGSP (National Glycohemoglobin Standardization Program) and the IFCC (International Federation of Clinical Chemistry and Laboratory Medicine).
Change in Pulse wave velocity | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the SphygmoCor system (AtCor Medical Pty Ltd Head Office, West Ryde, Australia).
Change in Fasting plasma glucose, apolipoproteins A1 and B, insulin ultrasensitive protein C and endothelial glycocalyx (syndecan-1, syndecan-4 and heparan sulfate proteins) | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the Abbott® Cobas 8000 Roche Diagnostics® system.
Change in Endothelial function | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the ENDO-PAT.
Change in 24-hour blood pressure | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the MAPA Mobil-O-graph.
Change in Educational level | At baseline of the 12 weeks intervention in the 2nd phase
  measured as the maximum level of education attained by each participant, classifying them as: cannot read or write, no studies, incomplete primary studies, primary studies, school graduate studies, higher baccalaureate studies, medium university studies, or higher university studies.
Change in Adherence to the Mediterranean diet | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  with the Mediterranean Diet Adherence Screener (MEDAS) questionnaire
Change in Sleep habits and quality of sleep | Baseline and at the end of the 12 weeks intervention in the 2nd and 3rd phase
  with the Pittsburgh Sleep Quality Index (PSQI)
Change in Comorbidities | At baseline of the 12 weeks intervention in the 2nd and 3rd phase
  with the Charlson comorbidity index.
Change in Attention | At baseline of the 12 weeks intervention in the 2nd and 3rd phase
  Using the Flanker Task test
Change in Working memory | At baseline of the 12 weeks intervention in the 2nd and 3rd phase
  Using the AWMA (Automated Working Memory Assessment) test
Change in Cognitive flexibility | At baseline of the 12 weeks intervention in the 2nd and 3rd phase
  Using the DCCS (Dimension Change Card Sort) test
Change in radial augmentation rate (rAIx) | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the SphygmoCor system (AtCor Medical Pty Ltd Head Office, West Ryde, Australia).
Change in central augmentation rate (cAIx) | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the SphygmoCor system (AtCor Medical Pty Ltd Head Office, West Ryde, Australia).
apolipoproteins A1 and B | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the Abbott® Cobas 8000 Roche Diagnostics® system.
insulin ultrasensitive protein C | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the Abbott® Cobas 8000 Roche Diagnostics® system.
endothelial glycocalyx (syndecan-1, syndecan-4 and heparan sulfate proteins) | Baseline and at the end of the 12 weeks intervention in the 2nd phase
  with the Abbott® Cobas 8000 Roche Diagnostics® system.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alvarez-Bueno C, Luceron-Lucas-Torres M, Ruiz-Hermosa A, Sequi-Dominguez I, Venegas-Sanabria LC, Medrano-Echeverria M, Visier-Alfonso ME, Rodriguez-Martin B. Protocol of the MOVI-ageing randomized controlled trial: a home-based e-Health intervention of cognitively demanding exercise for the improvement of cardiorespiratory fitness and cognitive function in older individuals. Front Public Health. 2023 Dec 22;11:1298316. doi: 10.3389/fpubh.2023.1298316. eCollection 2023. PMID 38186705